CLINICAL TRIAL: NCT02366299
Title: Comparison of Sedative Effects of Dexmedetomidine and Propofol on the Clinical Course of Delirium and Neuroinflammation in Patients With SIRS.
Brief Title: Comparison of Dexmedetomidine and Propofol on the Delirium and Neuroinflammation in Patients With SIRS.
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Moscow Regional Research and Clinical Institute (MONIKI) (Other Government)
Responsible Party: Principal Investigator, Valery V. Likhvantsev, Professor, senior researcher, Moscow Regional Research and Clinical Institute (MONIKI)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D-P-SIRS-220115
Record Dates: First submitted 2015-01-26; First posted 2015-02-19 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium | interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- dexmedetomidine (Active Comparator): Treatment of delirium by dexmedetomidine i.v. infusion
  Interventions: Drug: Dexmedetomidine
- propofol (Active Comparator): Treatment of delirium by propofol i.v. infusion
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Dexmedetomidine — Treatment of delirium by dexmedetomidine i.v. infusion
  Other Names: Dexdor
  Arms: dexmedetomidine
Drug: Propofol — Treatment of delirium by Propofol i.v. infusion
  Other Names: Diprivan
  Arms: propofol

SUMMARY:
Assessment of sedative effects of dexmedetomidine and propofol on the clinical course of delirium and neuroinflammation in patients with SIRS using CAM-ICU scale and protein S100b in serum.

ELIGIBILITY:
Inclusion Criteria:

* presence of delirium

Exclusion Criteria:

* presence of Alzheimer's disease
* any mental disorder
* presence of cancer

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-02; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
CAM-ICU scale | up to 5 days